CLINICAL TRIAL: NCT07214870
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NNC4005-0001 in Adults
Brief Title: A Research Study of a Potential New Medicine (NNC4005-0001) for Liver Disease in Adult Participants With Increased Body Weight and Liver Fat
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN4005-8221; UTN (Other: U1111-1319-8000)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC4005-0001 (Experimental): Participants will receive a single dose of NNC4005-0001 injected subcutaneously. Trial will include up to 6 ascending single-dose cohorts.
  Interventions: Drug: NNC4005-001
- Placebo (Placebo Comparator): Participants in each cohort will receive placebo matched to NNC4005-0001 injected subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC4005-001 — NNC4005-0001 will be given as a single ascending dose via subcutaneous route
  Arms: NNC4005-0001
Drug: Placebo — Placebo matched to NNC4005-0001 will be given via subcutaneous route
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to find out if NNC4005-0001 is well-tolerated and safe for people who have increased body weight and increased liver fat. Participants will receive either NNC4005-0001, which is the treatment being tested, or a placebo, which is a treatment that contains no active medicine. The study will last for about for about 7 to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-69 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) of 27.0-40.0 kilogram per square meter (kg/m^2) (both inclusive) at screening process.
* Hepatic fat fraction greater than or equal to (≥) 8% by magnetic resonance imaging proton density fat fraction (MRI-PDFF) within 17 days prior to dosing.
* No prior or present clinical history of metabolic dysfunction-associated steatohepatitis (MASH) diagnosis.

Exclusion criteria:

* Any condition, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Previous or current use of therapies for MASH or antifibrotic therapies (authorised or within aclinical trial).
* Use of high-dose vitamin E [greater than (>) 800 international unit (IU) per day], glucagon-like peptide-1 (GLP-1) agonists (such as liraglutide, dulaglutide, or semaglutide), glucose-dependent insulinotropic polypeptide (GIP)/GLP-1 agonists (such as tirzepatide), or pioglitazone within 6 months prior to screening.
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) levels greater than or equal (≥) 1.5× Upper Limit of Normal (ULN) at screening.
* Total bilirubin levels > 1.5 times ULN if direct bilirubin is within Normal Limits (WNL) at screening.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-05-14 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-emergent adverse event (TEAEs) | From dosing (day 1) until compeletion of end of study (EOS) visit on day 169
  Measured as count of events

SECONDARY OUTCOMES:
AUC(0-last): The area under the NNC4005-0001 plasma concentration-time curve from time zero to last measurable concentration after a single dose | From dosing (day 1) to 48 hours post-dose
  microgram*hour per milliliter (μg*h/mL)
Cmax: The maximum concentration of NNC4005-0001 in plasma | From dosing (day 1) to 48 hours post-dose
  Measured in microgram per millilitre
tmax: The time from dose administration to the maximum plasma concentration of NNC4005-0001 | From dosing (day 1) to 48 hours post-dose
  Hour
t1/2: Half life | From dosing (day 1) to 48 hours post-dose
  Hour
CLr: Renal clearance | From dosing (day 1) to 48 hours post-dose
  Liter/hour (L/h)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency' (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical Company, Inc, Montreal, Quebec, Canada